CLINICAL TRIAL: NCT03594149
Title: Efficiency of Antibacterial Prophylaxis (Levofloxacin) in Azacitidine Treated Patients
Brief Title: Efficiency of Antibacterial Prophylaxis in Azacitidine Treated Patients
Acronym: AZABAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHB 17.01
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
Keywords: levofloxacin, antibacterial prophylaxis, febrile episode
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antibacterial prophylaxis (Experimental): Levofloxacin 500 mg/d p.o. during the first 3 cycles of azacytidine
  Interventions: Drug: Levofloxacin
- control (No Intervention): No levofloxacin will be given.

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin 500 mg/d p.o.
  Other Names: LVF
  Arms: antibacterial prophylaxis

SUMMARY:
Infections are a major life-threatening complication in patients with myelodysplastic syndrome (MDS) or acute myeloid leukaemia (AML). Currently there is no guidelines about antibacterial prophylaxis to prevent infections in patients with myelodysplastic syndrome or acute myeloid leukaemia. The investigators will conduct a randomized prospective study to evaluate the benefit of prophylactic antibacterial by levofloxacin on febrile episode in Azacytidine treated patients (MDS and AML).

DETAILED DESCRIPTION:
This is a randomized prospective study with 2 arms to evaluate the efficacy of Levofloxacin prophylaxis in Azacytidine treated patients (MDS and AML) Levofloxacin will be given 500mg/d p.o. for the first three cycles of Azacytidine in patients randomized in arm antibacterial prophylaxis. In control arm patients will not received levofloxacin.

The expected duration of subject participation is one year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 18 years old
* SMD or AML treated with azacytidine (not previously treated)
* Life expectancy more than 3 months
* Performance status inferior to 3
* signed inform consent

Exclusion Criteria:

* allergy to quinolone
* previous event of tendopathy due to quinolone
* previous epileptic event
* systemic antibacterial prophylaxis the month before enrolment
* HIV positive
* bacterious infection of indetermined fever
* participation to an investigational drug trial
* Abnormalities in hepatic assessment
* QTc superior to 450 ms
* Pregnant or lactating women
* Myasthenia
* G6PD deficient
* severe and uncontrolled diabetes
* patient not able to understand trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Febrile episode occurrence | 3 cycles of 28 days
  Febrile episode occurrence during the3 first cycles of azacytidine requiring hospitalization and introduction of an antibiotic (with or without levofloxacin discontinuation

SECONDARY OUTCOMES:
one-year overall survival rate | one year
  overall survival at one year in both two arms
infectious agents documented in each arm | one year
  index of infectious agents in both two arms
infectious events rate | one year
  number of infectious events in both two arms
apparition of multi-drug resistant bacteria | one year
  index of multi-drug resistant bacteria in both two arms
duration of hospitalization | one year
  number of days of hospitalization and number of days of antibiotic or antifungal treatment
carbapenem and glycopeptide consumption in both two arms | 3 years
  consumption of carbapenem and glycopeptide during inclusion period and comparison with the 3 previous years
death causes | one year
  index of death causes in each arms
toxicity profile (adverse event) | one year
  toxicity will be established with description of adverse event in both two arms

CONTACTS AND LOCATIONS:
Overall Officials: Stamatoullas-Bastard Aspasia, MD, Principal Investigator — Centre Henri Becquerel
Locations (4):
- France (4):
  - CHU Amiens, Amiens
  - CHU Caen, Caen
  - CHRU Lille, Lille
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No